CLINICAL TRIAL: NCT04189757
Title: A Phase II Study of Acalabrutinib in Ibrutinib-Intolerant Mantle Cell Lymphoma
Brief Title: Acalabrutinib for the Treatment of Ibrutinib-Intolerant Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0421; NCI-2019-07927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0421 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib) (Experimental): Patients receive acalabrutinib PO BID on days 1-28. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence

SUMMARY:
This phase II trial studies how well acalabrutinib works in treating patients with mantle cell lymphoma that cannot tolerate ibrutinib. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the overall response rate (ORR) at the end of 3 cycles of acalabrutinib.

SECONDARY OBJECTIVES:

I. To assess the proportion of patients that are progression free without any of the following toxicities at the end of 3 cycles:

Ia. Recurrence of intolerable toxicities previously noted on ibrutinib. Ib. The occurrence of intolerable toxicities related to acalabrutinib defined as: grade 4 neutropenia or thrombocytopenia lasting greater than 7 days or any grade >= 3 non-hematologic toxicity as assessed by the investigator to be related to study drug).

II. To determine the efficacy of acalabrutinib, progression free survival (PFS) and duration of response (DOR) in patients.

III. To assess the safety profile of acalabrutinib in patient's intolerant to ibrutinib.

EXPLORATORY OBJECTIVE:

I. Sequential peripheral blood (PB)/plasma/tissue fine-needle aspiration (FNA) will be stored for evaluation of:

Ia. Clonal evolution with targeted sequencing (seq) and/or whole exome sequencing (WES) in sequential samples.

Ib. Pattern of mutation changes with acalabrutinib. Ic. Response predictors - mutations, cytokine-chemokines. Id. Minimal residual disease (MRD) assay using flow cytometry (FC) and circulating tumor-derived deoxyribonucleic acid (ctDNA) analysis.

Ie. Sequential immunologic studies with cytokines/chemokines, T cells and immunoglobulins.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 1 years, then annually for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mantle cell lymphoma with CD20 positivity and chromosome translocation t(11;14), (q13;q32) and/or overexpress cyclin D1 in tissue biopsy
* Include patients who require treatment (versus watch/wait)
* Prior treatment with ibrutinib discontinued for reasons other than progression
* Ibrutinib intolerance is defined as unacceptable toxicity where, in the opinion of the investigator, treatment should be discontinued in spite of optimal supportive care as a result of one of the following:

  * 2 or more grade >= 2 non-hematological toxicities; OR
  * 1 or more grade 3 >= 3 non-hematological toxicity; OR
  * 1 or more grade 3 neutropenia with infection or fever; OR,
  * Grade 4 hematologic toxicity which persists to the point that the investigator chose to stop therapy due to toxicity NOT progression

    * Toxicity must have resolved to =< grade 1 prior to acalabrutinib dosing
* Understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form
* Bi-dimensional measurable disease using the Cheson criteria (measurable disease by positron emission tomography [PET]-computed tomography [CT] scan defined as at least 1 lesion that measures >= 1.5 cm in single dimension). Gastrointestinal, bone marrow or spleen only patients are allowable
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Absolute neutrophil count (ANC) > 1,000/mm^3

  * Patients who have bone marrow infiltration by mantle cell lymphoma (MCL) are eligible if their ANC is >= 500/mm^3 (growth factor allowed) or their platelet level is equal to or > 20,000/mm^3. These patients should be discussed with either the principal investigator (PI) or co-PI of the study for final approval
* Platelet count > 75,000/mm^3

  * Patients who have bone marrow infiltration by MCL are eligible if their ANC is >= 500/mm^3 (growth factor allowed) or their platelet level is equal to or > 20,000/mm^3. These patients should be discussed with either the PI or co-PI of the study for final approval
* Serum bilirubin < 1.5 mg/dl
* Creatinine (Cr) clearance minimum to 30 mL/min per the Cockcroft-Gault formula as acalabrutinib pharmacokinetic (PK) has not been evaluated in patients with severe renal impairment (estimated glomerular filtration rate [eGFR] < 29 mL/min/1.7 3^m2, MDRD) or renal impairment requiring dialysis
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. Gilbert's disease is allowed
* Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated with life expectancy of > 3 years. PI can use clinical judgement in the best interest of patients
* Women of childbearing potential (WOBP) must have a negative serum or urine pregnancy test. WOBP and males must be willing to use highly effective methods of birth control prior to starting therapy. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for one week after the last dose of acalabrutinib. For male subjects with a pregnant or non-pregnant WOCBP partner, should use barrier contraception even if they have had a successful vasectomy
* Patients who were not placed originally on ibrutinib by the providers due to concerns for worsening of comorbidities due to ibrutinib, such as atrial fibrillation can be included after cardiology clearance
* Patients with well-controlled human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS) would be eligible

Exclusion Criteria:

* Prior treatment with acalabrutinib
* History of BTK mutations conferring resistance to BTK inhibitors. Known mutations in the BTK gene that confer resistance to ibrutinib in mantle cell lymphoma include (e.g. BTK C481S, C481R mutations)
* Progressive disease while on ibrutinib therapy. Patients who progressed while on ibrutinib therapy will be excluded from the study, patients who discontinue ibrutinib due to anaphylaxis or hypersensitivity reaction related to ibrutinib will be excluded from participation in the study
* Known history of drug-specific hypersensitivity or anaphylaxis to ibrutinib (including active product or excipient components)
* Pregnant or breast-feeding females
* Patients with active hepatitis B infection. Those with prior hepatitis (hep)-B vaccination (i.e., anti-HBs antibody positive) or natural immunity as evidenced by the presence of anti-HBs and anti-HBc positivity are eligible to enroll. (Known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal [GI] consultation)
* Patients with central nervous system involvement with mantle cell lymphoma or with suspected or confirmed progressive multifocal leukoencephalopathy (PML) are excluded since those patients have very poor prognosis, need aggressive intensive chemoimmunotherapy and intrathecal chemotherapy along with BTK inhibitors and these patients would not be eligible for single agent acalabrutinib as proposed in this study
* Active bleeding, history of bleeding diathesis (such as hemophilia or Von-Willebrand disease), Any history of intracranial bleed or stroke within 6 months of first dose of study drug
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Ongoing adverse events from prior ibrutinib therapy (except persistent hematologic toxicity if meeting entry criteria). The PI should determine if AEs are an ongoing sequel of prior BTK therapy such as fungal infections, skin rash, diarrhea, fatigue, cramps and colitis or if the patient has resolved AE and is free of these adverse events >= 2 months after stopping ibrutinib)
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of acalabrutinib
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before first dose of study drug
* Major surgery within 4 weeks of initiation of therapy
* Requires anticoagulation with warfarin or equivalent vitamin K antagonist
* Concomitant use of corticosteroids at > 10 mg prednisone or equivalent per day
* Requires treatment with strong CYP3A inhibitors or inducers
* Any of the following cardiac related conditions:

  * New York Heart Association (NYHA) class III and IV heart failure,
  * Active/symptomatic coronary artery disease,
  * Myocardial infarction in the preceding 6 months,
  * Significant conduction abnormalities, including but not limited to:

    * Left bundle branch block,
    * 2nd degree atrioventricular (AV) block type II,
    * 3rd degree block,
    * QT prolongation (corrected QT interval [QTc] > 500 msec),
    * Sick sinus syndrome,
    * Ventricular tachycardia,
    * Symptomatic bradycardia (heart rate < 50 bpm),
    * Persistent and uncontrolled atrial fibrillation.
  * Uncontrolled hypertension,
  * Hypotension,
  * Light headedness and syncope
* Acute infection requiring systemic anti-microbial treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to initiation of therapy
* Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole or pantoprazole). Subjects receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
* Any other serious medical condition including, but not limited to, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease (COPD), renal failure, psychiatric illness or social circumstances that, in the investigator's opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form or complying with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (complete response + partial response) | At the end of cycle 3 (each cycle is 28 days)
  The primary end point will be met if > 50% patients attain response (half of patients responding without intolerance). Logistic regression may be utilized to assess the effect of patient prognostic factors on the response rate. Intent-to-treat analysis will be applied to the eligible patients.

SECONDARY OUTCOMES:
Incidence of adverse events | At the end of cycle 3 (each cycle is 28 days)
  Logistic regression may be utilized to assess the effect of patient prognostic factors on the incidence of adverse events. Toxicity and safety data will be summarized by frequency tables for all patients and then will be reviewed for relatedness to acalabrutinib. Per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received. Also, time to event and time to event resolution will be calculated.
Progression free survival | Up to 6 years
  The distribution of time-to-event endpoints including progression free survival will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Overall survival | Up to 6 years
  The distribution of time-to-event endpoints including overall survival will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Preetesh Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04189757/ICF_000.pdf